CLINICAL TRIAL: NCT06844136
Title: ChemoINTEL Assay Algorithm Development Study: In-Vitro Cytotoxic Drug Induced Apoptosis Correlation with Patient Clinical Response to Administered Chemotherapy in Patients with Advanced Stage Epithelial Ovarian Cancer.
Brief Title: ChemoINTEL Assay Algorithm Development Study: In-Vitro Cytotoxic Drug Induced Apoptosis Correlation with Patient Clinical Response to Administered Chemotherapy in Patients
Acronym: ChemoINtel
Status: Recruiting | Type: Observational
Sponsor: Pierian Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 201600013
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour Biopsy Blood sample Ascites fluids
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: De Novo (no prior cytotoxic therapy) receiving primary cytoreductive surgery and adjuvant chemotherapy
  Interventions: Other: No intervention
- Group 2: De Novo (no prior cytotoxic therapy) receiving neoadjuvant chemotherapy and interval cytoreductive surgery followed by additional chemotherapy
  Interventions: Other: No intervention
- Group 3: Recurrent (one or more prior lines of previous cytotoxic therapy) receiving next line of chemotherapy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a prospective, non-randomized, observational, clinical development study. Pierian Biosciences is utilizing ChemoINTEL and ImmunoINTEL assay measurements in human tumour cells from patients with advanced stage epithelial ovarian cancer (EOC) to develop a mathematical algorithm which will be able to predict a patient's tumour's sensitivity to specific chemotherapy drugs. The study involves using a sample of tumour biopsy taken during standard of care surgery, with a matched blood sample if possible. Medical history, pathology information and information on chemotherapy for up to 6 cycles will be requested. The information will then be used to developed an algorithm to predict tumour sensitivity to treatment.

DETAILED DESCRIPTION:
The justification for this study is to provide evidence based predictive scoring of available cytotoxic drug based on the patient's own tumour response characteristics to guide the physician's therapeutic selections and enable a personalized treatment plan. This study will generate a predictive algorithm using individual patient tumour ChemoINTEL and ImmunoINTEL assay response metrics paired with the patient's clinical response data. Subsequent Clinical Validation and Clinical Utility Studies will be conducted to provide further evidence for utilization of personalized predictive response scoring of available therapeutics enabling section of personalized treatment regiments based on each patient's unique tumour as an improvement over guideline driven approaches.

Cancer treatments and selection of cytotoxic drugs used in different situations continues to be guideline driven. These selections are generally based on treatment protocols developed as a result of large, population-based, prospective, randomized, multicenter, well-controlled phase 3 studies that analyze treatment outcomes (progression-free survival [PFS] and overall survival [OS]) as a function of treatment received by patient cohorts. This approach was necessitated by the stark reality that no "predictive" or "treatment-directing" diagnostic technologies were available, a circumstance that, to an overwhelming degree, remains unaltered. Treatment "guidelines" are utilized by most oncologists globally as they recommend treatment algorithms and options based on data with the highest levels of evidence. Several treatment guidelines are available globally such as those produced by the National Comprehensive Cancer Network (NCCN), the American Society of Clinical Oncology (ASCO), and European Society of Medical Oncology (ESMO). These guidelines provide evidence-based recommendations to guide physicians and outline appropriate methods of treatment and care. The guidelines often address specific clinical situations (disease oriented) on the use of approved medical products, procedures, or tests (modality oriented).

ELIGIBILITY:
Screening Criteria:

* Females ≥18 years of age
* Patient must sign an Informed Consent Form
* Patient is suspected to have one of the following

  * advanced stage Epithelial Ovarian Cancer (EOC)
  * advanced stage Primary Peritoneal Carcinomatosis
  * advanced stage Fallopian Tube Carcinoma

Inclusion Criteria:

* Females ≥18 years of age
* Diagnosis by pathology of one of either advanced stage EOC, Primary Peritoneal Carcinomatosis, or Fallopian Tube Carcinoma

  * Newly diagnosed
  * Recurrent
* Patient provided an evaluable tumor or peritoneal fluid specimen prior to initiating chemotherapy for ChemoINTEL assay analysis
* Patient received at least 3 cycles of standard of care chemotherapy for advanced stage EOC with single agent or combination of drugs summarised as below, following biopsy OR surgical resection

  * Carboplatin
  * Cisplatin
  * Cyclophosphamide-4HC active metabolite
  * Docetaxel
  * Doxorubicin
  * Etoposide
  * Fluorouracil
  * Gemcitabine
  * Ifosfamide-4HI active metabolite
  * Irinotecan
  * Oxaliplatin
  * Paclitaxel
  * Pemetrexed
  * Topotecan
  * Vinorelbine
  * Bevacizumab (Avastin)
* Patients will have an appropriate evaluation after their third cycle and sixth cycle of SOC chemotherapy to document response by either RECIST 2009 v1.1, CA-125 KELIM Scoring, and/or circulating tumor DNA longitudinal monitoring
* Patient signed Informed Consent Form

Exclusion Criteria:

* Patient has not signed an ICF to participate in a clinical investigation
* Patient has a cancer other than advanced stage EOC
* Patient did NOT receive SOC chemotherapy, single agents or combination treatment from the indicated list above.
* Patients did NOT have sufficient viable cells recovered from either a fresh tumor dissociation or peritoneal fluid specimen collected prior to initiating chemotherapy available for the minimum ChemoINTEL assay analysis of Carboplatin, Cisplatin, Docetaxel, and Paclitaxel test conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with ovarian cancer
Study Population: Ovarian cancer diagnosis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Prediction Algorithm | 2 years
  To develop a prediction algorithm that uses input from the ChemoINTEL and ImmunoINTEL assay metric results and provides an accurate prediction of a patient's cancer's sensitivity to specific chemotherapeutic agents by assessing the patient's response based on either RECIST criteria (v 1.1, 2009), CA-125 KELIM Score, and/or circulating tumor DNA changes to the administered chemotherapy following three cycles of SOC chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Henry, Study Director — Pierian Biosciences Ltd
Locations (1):
- Liverpool Women's NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Plan to disseminate the findings and publish the findings, all data will be anonymised